CLINICAL TRIAL: NCT03881852
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, 3-Week Crossover Study to Assess the Efficacy and Safety of AXS-12 in Subjects With Cataplexy and Excessive Daytime Sleepiness in Narcolepsy
Brief Title: Clinical Outcomes in Narcolepsy and Cataplexy: An Evaluation of Reboxetine Treatment (CONCERT)
Acronym: CONCERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AXS-12-201
Record Dates: First submitted 2019-03-15; First posted 2019-03-20 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Narcolepsy; Cataplexy Narcolepsy; Excessive Sleepiness
Keywords: CONCERT; AXS-12; EDS; Cataplexy; Narcolepsy; Axsome; Reboxetine
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence; Cataplexy | interventions — Reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-12 (reboxetine) (Experimental)
  Interventions: Drug: AXS-12 (Reboxetine)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-12 (Reboxetine) — Dosed orally, twice daily for up to 3 weeks
  Arms: AXS-12 (reboxetine)
Drug: Placebo — Dosed orally, twice daily for up to 3 weeks
  Arms: Placebo

SUMMARY:
CONCERT (Clinical Outcomes in Narcolepsy and Cataplexy: An Evaluation of Reboxetine Treatment) is a Phase 2, double-blind, randomized, placebo-controlled, crossover, multicenter trial of AXS-12 in patients with narcolepsy. Subjects meeting the entry criteria will be randomized in a 1:1 ratio either to placebo for three weeks followed by AXS-12 (up to 10 mg daily) for three weeks, or to AXS-12 (up to 10 mg daily) for three weeks followed by placebo for three weeks. Efficacy assessments will include the frequency of cataplexy attacks, and measures of other symptoms of narcolepsy.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects between 18 and 70 years of age, inclusive
* Primary diagnosis of narcolepsy with cataplexy
* Willing and able to comply with the study requirements

Exclusion Criteria:

* Other clinically significant conditions potentially causing EDS
* Clinically significant psychiatric disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - CONCERT Study Site, Birmingham, Alabama
  - CONCERT Study Site, Alameda, California
  - CONCERT Study Site, Santa Ana, California
  - CONCERT Study Site, Boulder, Colorado
  - CONCERT Study Site, Miami, Florida
  - CONCERT Study Site, St. Petersburg, Florida
  - CONCERT Study Site, Gainesville, Georgia
  - CONCERT Study Site, Fort Wayne, Indiana
  - CONCERT Study Site, Chevy Chase, Maryland
  - CONCERT Study Site, The Bronx, New York
  - CONCERT Study Site, Cincinnati, Ohio
  - CONCERT Study Site, Columbia, South Carolina
  - CONCERT Study Site, Austin, Texas
  - CONCERT Study Site, San Antonio, Texas

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Crossover Design: Subjects meeting the entry criteria will be randomized in a 1:1 ratio either to Sequence 1 [AXS-12 (up to 10 mg daily) for three weeks followed by placebo for three weeks] or Sequence 2 [placebo for three weeks followed by AXS-12 (up to 10 mg daily) for three weeks].
Groups:
- Sequence 1: Sequence 1 - AXS-12 (reboxetine) for three weeks followed by placebo for three weeks
- Sequence 2: Sequence 2 - Placebo for three weeks followed by AXS-12 (reboxetine) for three weeks
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2
Started | 11 | 10
Dosed With AXS-12 | 11 | 10
Dosed With Placebo | 10 | 10
Completed | 10 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (12.44) | 32.9 (6.74) | 32.6 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average Total Number of Cataplexy Attacks
Description: Presented as LSmeans. A positive change is indicative of improvement.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: weekly cataplexy attacks
Arm/Group | AXS-12 (Reboxetine) | Placebo
Number analyzed (Participants) | 21 | 20
weekly cataplexy attacks | 13.0 (3.5) | -0.28 (3.5)
Statistical Analysis 1: Comparison: AXS-12 (Reboxetine) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — P-value calculated from LSMean

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the randomization visit through 7 days after the last dosing date for non-serious AEs and 30 days after the last dosing for serious AEs.
Description: Safety Population includes all subjects who received study drug.
Groups:
- AXS-12 (Reboxetine): Adverse events collected while subjects were in the AXS-12 (reboxetine) period of either Sequence 1 or Sequence 2.
- Placebo: Adverse events collected while subjects were in the Placebo period of either Sequence 1 or Sequence 2.
Arm/Group | AXS-12 (Reboxetine) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 9/21 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-12 (Reboxetine) (N=21) | Placebo (N=20)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and SAP (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03881852/Prot_SAP_000.pdf
  • Statistical Analysis Plan: SAP only (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT03881852/SAP_001.pdf